CLINICAL TRIAL: NCT01074723
Title: Bioavailability of Added B-cryptoxanthin and Phytosterols; In Vitro and in Vivo Interactions and Effect on Bone Remodelling and Cardiovascular Risk Markers
Brief Title: B-cryptoxanthin and Phytosterols on Bone Remodeling and Cardiovascular Risk Factors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Fernando Granado Lorencio, Dr. Fernando Granado lorencio, Puerta de Hierro University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: AGL-2008-02591-C02-02
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Postmenopausal Disorder
Keywords: b-cryptoxanthin; cholesterol; bone markers; Osteoporosis; cardiovascular risk; post-menopausal women
MeSH Terms: conditions — Osteoporosis | interventions — Phytosterols; Carotenoids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- b-cryptoxanthin (Experimental)
  Interventions: Dietary Supplement: b-cryptoxanthin and phytosterols
- phytosterols (Experimental)
  Interventions: Dietary Supplement: b-cryptoxanthin and phytosterols
- b-cryptoxanthin plus phytosterols (Experimental)
  Interventions: Dietary Supplement: b-cryptoxanthin and phytosterols

INTERVENTIONS:
Dietary Supplement: b-cryptoxanthin and phytosterols — Fruit juices containing b-cryptoxanthin (ca. 1 mg), phytosterols (ca 1.7g) or both will be consumed for 4 weeks with a 4-week washout in between.
  Other Names: carotenoids, plant sterols

SUMMARY:
We, the investigators, aim to study, in vitro and in vivo, the bioavailability of added b-cryptoxanthin and phytosterols and evaluate in vivo its effect on biochemical markers of bone remodelling and cardiovascular risk. Specifically, we will 1) assess the stability in the food and the bioavailability of b-cryptoxanthin in the presence of phytosterols (absorption modifiers) by using a complementary approach; in vitro and in vivo studies; and 2) we will study in post-menopausal women (target group) the biological effect (bioefficacy) associated with the regular consumption of modified milk-based fruit beverages (containing b-cryptoxanthin and phytosterols) by assessing changes in biochemical markers of bone turnover and cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women, 45-60 years old

Exclusion Criteria:

* Dieting
* Food allergy (to any components provided)
* Hormone replacement therapy
* Cholesterol lowering drugs, antiresorptive or anabolic bone drugs
* Calcium and vitamin D supplements
* Soybean products
* Vitamin-mineral supplements
* Fibre supplements
* Commercially available enriched foods (i.e. w-3, phytosterols,carotenoids,...)

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Serum b-cryptoxanthin | 4 weeks

SECONDARY OUTCOMES:
Serum Cardiovascular risk markers | 4 weeks
Serum bone markers | 4 weeks
Genetic variability (polymorphisms)and DNA oxidative damage | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Puerta de Hierro University Hospital, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Granado-Lorencio F, de Las Heras L, Millan CS, Garcia-Lopez FJ, Blanco-Navarro I, Perez-Sacristan B, Dominguez G. beta-Cryptoxanthin modulates the response to phytosterols in post-menopausal women carrying NPC1L1 L272L and ABCG8 A632 V polymorphisms: an exploratory study. Genes Nutr. 2014 Sep;9(5):428. doi: 10.1007/s12263-014-0428-0. Epub 2014 Aug 28. PMID 25163590
- [Derived] Granado-Lorencio F, Lagarda MJ, Garcia-Lopez FJ, Sanchez-Siles LM, Blanco-Navarro I, Alegria A, Perez-Sacristan B, Garcia-Llatas G, Donoso-Navarro E, Silvestre-Mardomingo RA, Barbera R. Effect of beta-cryptoxanthin plus phytosterols on cardiovascular risk and bone turnover markers in post-menopausal women: a randomized crossover trial. Nutr Metab Cardiovasc Dis. 2014 Oct;24(10):1090-6. doi: 10.1016/j.numecd.2014.04.013. Epub 2014 May 6. PMID 24909799